CLINICAL TRIAL: NCT02555852
Title: Proton Pump Inhibitors and the Risk of Hospitalization for Community-acquired Pneumonia: Replicated Cohort Studies With Meta-analysis
Brief Title: Proton Pump Inhibitors and Risk of Community-acquired Pneumonia
Status: Completed | Type: Observational
Sponsor: Canadian Network for Observational Drug Effect Studies, CNODES (Other)
Collaborators: Drug Safety and Effectiveness Network, Canada (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: CNODES_DEMO-2
Record Dates: First submitted 2015-09-18; First posted 2015-09-22 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Gastroesophageal Reflux Disease (GERD); Community-acquired Pneumonia
Keywords: Proton Pump Inhibitors; Pneumonia; NSAIDs; Histamine H2 Antagonists; Drug safety
MeSH Terms: conditions — Gastroesophageal Reflux; Community-Acquired Pneumonia; Pneumonia | interventions — Esomeprazole; Proton Pump Inhibitors; Omeprazole; Pantoprazole; Lansoprazole; Rabeprazole; Cimetidine; Histamine H2 Antagonists; Ranitidine; Famotidine; Nizatidine; niperotidine; roxatidine acetate; ranitidine bismuth citrate; lafutidine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Users of PPIs: Exposure to proton pump inhibitors (PPIs) will be defined as a prescription for a PPI (esomeprazole, omeprazole, pantoprazole, lansoprazole, rabeprazole, and combinations) on the same day as the cohort entry defining prescription for an NSAID.
  Interventions: Drug: esomeprazole; Drug: omeprazole; Drug: pantoprazole; Drug: lansoprazole; Drug: rabeprazole
- Users of H2RAs: Exposure to histamine-2 receptor antagonists (H2RAs) will be defined as a prescription for a H2RA (cimetidine, ranitidine, famotidine, nizatidine, niperotidine, roxatidine, ranitidine bismuth citrate, lafutidine, cimetidine combinations, and famotidine combinations) on the same day as the cohort entry defining prescription for an NSAID.
  Interventions: Drug: cimetidine; Drug: ranitidine; Drug: famotidine; Drug: nizatidine; Drug: niperotidine; Drug: roxatidine; Drug: ranitidine bismuth citrate; Drug: lafutidine; Drug: cimetidine combinations; Drug: famotidine combinations
- Unexposed group (Reference): Patients that are considered to be unexposed will be defined as patients not prescribed a PPI or H2RA on the same day as the cohort entry defining prescription for an NSAID.

INTERVENTIONS:
Drug: esomeprazole — Exposure to esomeprazole (ATC A02BC05, B01AC56, M01AE52, A02BD06) will be defined as a prescription for esomeprazole on the same day as a ≥ 30 day NSAID prescription.
  Other Names: Proton pump inhibitor
  Groups: Users of PPIs
Drug: omeprazole — Exposure to omeprazole (ATC A02BC01, A02BD01) will be defined as a prescription for omeprazole on the same day as a ≥ 30 day NSAID prescription.
  Other Names: Proton pump inhibitor
  Groups: Users of PPIs
Drug: pantoprazole — Exposure to pantoprazole (ATC A02BC02, A02BD04) will be defined as a prescription for pantoprazole on the same day as a ≥ 30 day NSAID prescription.
  Other Names: Proton pump inhibitor
  Groups: Users of PPIs
Drug: lansoprazole — Exposure to lansoprazole (ATC A02BC03, A02BD07, A02BD03, A02BD02) will be defined as a prescription for lansoprazole on the same day as a ≥ 30 day NSAID prescription.
  Other Names: Proton pump inhibitor
  Groups: Users of PPIs
Drug: rabeprazole — Exposure to rabeprazole (ATC A02BC04) will be defined as a prescription for rabeprazole on the same day as a ≥ 30 day NSAID prescription.
  Other Names: Proton pump inhibitor
  Groups: Users of PPIs
Drug: cimetidine — Exposure to cimetidine (ATC A02BA01) will be defined as a prescription for cimetidine on the same day as a ≥ 30 day NSAID prescription.
  Other Names: histamine-2 receptor antagonist
  Groups: Users of H2RAs
Drug: ranitidine — Exposure to ranitidine (A02BA02) will be defined as a prescription for ranitidine on the same day as a ≥ 30 day NSAID prescription.
  Other Names: histamine-2 receptor antagonist
  Groups: Users of H2RAs
Drug: famotidine — Exposure to famotidine (A02BA03) will be defined as a prescription for famotidine on the same day as a ≥30 day NSAID prescription.
  Other Names: histamine-2 receptor antagonist
  Groups: Users of H2RAs
Drug: nizatidine — Exposure to nizatidine (A02BA04) will be defined as a prescription for nizatidine on the same day as a ≥ 30 day NSAID prescription.
  Other Names: histamine-2 receptor antagonist
  Groups: Users of H2RAs
Drug: niperotidine — Exposure to niperotidine (A02BA05) will be defined as a prescription for niperotidine on the same day as a ≥ 30 day NSAID prescription.
  Other Names: histamine-2 receptor antagonist
  Groups: Users of H2RAs
Drug: roxatidine — Exposure to roxatidine (A02BA06) will be defined as a prescription for roxatidine on the same day as a ≥ 30 day NSAID prescription.
  Other Names: histamine-2 receptor antagonist
  Groups: Users of H2RAs
Drug: ranitidine bismuth citrate — Exposure to ranitidine bismuth citrate (A02BA07) will be defined as a prescription for ranitidine bismuth citrate on the same day as a ≥ 30 day NSAID prescription.
  Other Names: histamine-2 receptor antagonist
  Groups: Users of H2RAs
Drug: lafutidine — Exposure to lafutidine (A02BA08) will be defined as a prescription for lafutidine on the same day as a ≥ 30 day NSAID prescription.
  Other Names: histamine-2 receptor antagonist
  Groups: Users of H2RAs
Drug: cimetidine combinations — Exposure to cimetidine combinations (A02BA51) will be defined as a prescription for cimetidine combinations on the same day as a ≥ 30 day NSAID prescription.
  Other Names: histamine-2 receptor antagonist
  Groups: Users of H2RAs
Drug: famotidine combinations — Exposure to famotidine combinations (A02BA53) will be defined as a prescription for famotidine combinations on the same day as a ≥ 30 day NSAID prescription.
  Other Names: histamine-2 receptor antagonist
  Groups: Users of H2RAs

SUMMARY:
The purpose of the study is to determine whether proton pump inhibitors (PPIs), a medication used to treat gastric conditions, increase the risk of hospitalization for community-acquired pneumonia (HCAP).

The investigators will carry out separate population-based cohort studies using administrative health databases in eight jurisdictions in Canada, the US, and the UK. Cohort entry will be defined by the initiation of an oral non-steroidal anti-inflammatory drug, with follow-up until hospitalization for pneumonia or end of follow-up (6 months). The results from the separate sites will be combined using a statistical approach called meta-analysis to provide an overall assessment of the risk of HCAP with PPIs.

DETAILED DESCRIPTION:
Previous observational studies have found an association between proton pump inhibitors (PPIs), a class of medications used to treat gastric conditions, and the risk of community acquired pneumonia. These studies, however, had important limitations including confounding by indication and protopathic bias. The purpose of this study is to determine whether PPIs increase the risk of hospitalization for community-acquired pneumonia (HCAP). To overcome the limitations of previous studies that examined this issue, this study will be conducted in a cohort of new users of non-steroidal anti-inflammatory drugs (NSAIDs), in whom PPIs are often prescribed prophylactically to prevent dyspepsia and other gastric side effects.

The investigators will use a common-protocol approach to conduct retrospective cohort studies using administrative health care data from eight jurisdictions (the Canadian provinces of Alberta, Saskatchewan, Manitoba, Ontario, Quebec, and Nova Scotia, as well as the United States (US) MarketScan, and the United Kingdom (UK) General Practice Research Database [GPRD]). Briefly, the Canadian databases include population-level data on physician billing, diagnoses and procedures from hospital discharge abstracts, and dispensations for prescription drugs. Alberta, Nova Scotia, Ontario, and Quebec data will be restricted to patients aged 65 years and older as prescription data are not available for younger patients. For Quebec, a 10% random sample of eligible patients will be used. The GPRD is a clinical database that is representative of the UK population and contains the records for patients seen at over 680 general practitioner practices in the UK. US MarketScan includes individuals and their dependents covered by large U.S. employer health insurance plans, and government and public organizations. As Medicare eligibility begins for those above the age of 65, the US MarketScan data will be restricted to patients aged 40 to 65 years in order to ensure complete data capture.

In each jurisdiction, the investigators will assemble a source population that includes all patients with a prescription for an oral NSAID (WHO Anatomical Therapeutic Chemical (ATC) Code M01A). From this source population, a study cohort will be created including all patients who received a prescription for an oral NSAID of ≥ 30 days duration, as patients receiving short duration prescriptions are unlikely to be prescribed a PPI for prophylactic reasons. The date of prescription (for the GPRD) or dispensation (for all other sites) of the oral NSAID will define the date of study cohort entry.

Patients will be followed from the date of study cohort entry until an event (defined below) or censoring due to death, departure from the database, end of follow-up (180 days), or the end of the study period (September 30, 2011 or the last date of data availability at that site), whichever occurs first. Patients will be permitted to enter the cohort multiple times provided that all inclusion criteria are met.

The investigators will create three mutually exclusive exposure categories: 1) PPI users, 2) H2RA users, and 3) unexposed patients. The investigators will use an analysis analogous to an intention-to-treat approach. Exposure to PPIs will be defined as a prescription for a PPI (esomeprazole, omeprazole, pantoprazole, lansoprazole, rabeprazole) on the same day as their cohort entry defining prescription for an NSAID. Exposure to H2RAs will be defined as a prescription for a H2RA (cimetidine, ranitidine, famotidine, nizatidine, niperotidine, roxatidine, ranitidine bismuth citrate, lafutidine, cimetidine combinations, and famotidine combinations) on the same day as their cohort entry defining prescription for an NSAID. Patients that are considered to be unexposed will be defined as patients not prescribed a PPI or H2RA on the same day as their cohort entry defining prescription for an NSAID. The primary outcome will be defined as incident HCAP during the 6 months following initiation of NSAID therapy.

Multiple logistic regression will be used to estimate site-specific adjusted odds ratios (aORs) and corresponding 95% confidence intervals (CIs) for the association of incident HCAP at 6 months and PPI exposure. This is considered the primary analysis. Several sensitivity analyses will be performed to assess the robustness of study results. Such analyses include: restricting analyses to a single, random, observation per patient; excluding patients who received a prescription for a PPI, H2RA, or NSAID in the 12 months before cohort entry; and excluding crossovers between PPI and H2RAs. High dimensional propensity scores will be estimated for all patients in the cohort using logistic regression. Finally, all site-specific estimates will be meta-analyzed using fixed models with inverse variance weighting. The amount of between-site heterogeneity will be estimated using the I-squared statistic.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a first oral NSAID prescription
* Patients at least 40 years of age (except Alberta, Ontario, and Nova Scotia, where patients will be at least 66 years of age)
* Patients with at least 1 year of history in the database.

Exclusion Criteria:

* Patients aged < 40 years at cohort entry (or < 66 in Alberta, Ontario, and Nova Scotia)
* Received a prescription for a PPI, a H2RA, or a NSAID (any route of administration) in the 6 months prior to cohort entry
* Had an HCAP (ICD-9-CM code (in any field): 480.x-487.x; ICD-10-CA code: J10.0 - J18.9) or an extended emergency room visit for community-acquired pneumonia in the year prior to cohort entry (where available)
* Hospitalized at the time of cohort entry
* Received a prescription for medications used for the treatment of tuberculosis (ATC Code J04A) (where available)
* Had a history of cancer (other than non-melanoma skin cancer) in the year prior to cohort entry
* Hospitalized >3 days within the 30 days before cohort entry
* Had <1 year of continuous observation time in the database prior to cohort entry

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In each jurisdiction, the investigators will assemble a study cohort that includes all patients with a new prescription for an oral NSAID between January 1, 1997 and March 31, 2010. The date of study cohort entry is defined by the prescription date of the newly-prescribed NSAID.
Sampling Method: Probability Sample
Enrollment: 4238504 (Actual)
Dates: Start 2011-09; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Hospitalization for Community-Acquired Pneumonia (HCAP) | Patients will be followed from the date of study cohort entry until HCAP, censoring, or for up to 6 months.
  HCAP during the 6 months following cohort entry
  Patients with HCAP with any of the following diagnostic codes: ICD-9: 487.0, 487.1, 487.0, 487.1, 487.0, 480.9, 481.x, 482.2, 482.0, 482.1, 482.30, 482.31, 482.32, 482.39, 482.40, 482.41, 482.42, 482.49, 482.81, 482.82, 482.83, 482.89, 482.9, 483.0, 484.7, 484.8, 485.X, 481.X, 486.X ; ICD-10: J10.0, J11.0, J11.1, J12.9, J13, J14, J15.X, J16.8, J17.0, J17.2, J17.3, J17.8, J18.0, J18.1, J18.8, J18.9.

CONTACTS AND LOCATIONS:
Overall Officials: Kristian Filion, PhD, Principal Investigator — Lady Davis Institute for Medical Research, Jewish General Hospital - McGill University
Locations (1):
- Lady Davis Institute for Medical Research, Jewish General Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Result] Filion KB, Chateau D, Targownik LE, Gershon A, Durand M, Tamim H, Teare GF, Ravani P, Ernst P, Dormuth CR; CNODES Investigators. Proton pump inhibitors and the risk of hospitalisation for community-acquired pneumonia: replicated cohort studies with meta-analysis. Gut. 2014 Apr;63(4):552-8. doi: 10.1136/gutjnl-2013-304738. Epub 2013 Jul 15. PMID 23856153
- See also: This organization's website describing general functions, other CNODES projects, and investigator profiles. — http://www.cnodes.ca